CLINICAL TRIAL: NCT05191212
Title: Real-time Lymphatic Channel Visualization Compared With Conventional Cervical Indocyanine Green Injection for Sentinel Lymph Node Mapping in Early-stage Endometrial Cancer
Brief Title: Real-time Lymphatic Channel Visualization Improves Bilateral Sentinel Lymph Node Detection in Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Gokhan Demirayak, MD, Assoc. Professor of Gynecologic Oncology, University of Health Sciences, Bakırköy Dr. Sadi Konuk Training and Research Hospital, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021/455
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Endometrial Cancer; Endometrial Neoplasms; Sentinel Lymph Node Biopsy (SLNB)
Keywords: Endometrial cancer; Sentinel lymph node; İndocyanine green; Lymphatic channel; Lymphatic Channel Visualization; Uterine cancer; Da Vinci Surgical System; Robotic Surgery; Real-time Visualization; Fluorescence Imaging; Near-Infrared Fluorescence; Gynecologic Oncology; Endometrial neoplasms
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, parallel-group study in which patients with clinical early-stage endometrial cancer are assigned to either conventional cervical indocyanine green (ICG) injection or real-time lymphatic channel-guided ICG injection for sentinel lymph node mapping. Each participant undergoes only one technique according to randomization.
Masking Description: Not applicable. This is an open-label surgical trial; no parties were masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental injection (Experimental): Cervical indocyanine green injections until real-time visualization of the afferent lymphatic channels bilaterally.
  Interventions: Procedure: indocyanine green
- Standart injection (Active Comparator): Cervical indocyanine green injections group
  Interventions: Procedure: indocyanine green

INTERVENTIONS:
Procedure: indocyanine green — Cervical indocyanine green injection for the detection of sentinel lymph node

SUMMARY:
Endometrial cancer is the most common malignancy of the female genital tract. Standard treatment for early-stage disease includes hysterectomy, bilateral salpingo-oophorectomy, and lymph node assessment. Sentinel lymph node (SLN) mapping with indocyanine green (ICG) has become widely used as an alternative to systematic lymphadenectomy due to lower morbidity and high detection rates.

This randomized clinical trial was designed to compare conventional cervical ICG injection with a modified technique, in which injection is continued until real-time lymphatic channels are visualized intraoperatively, for bilateral SLN detection in patients with clinical early-stage endometrial cancer undergoing robotic surgery.

DETAILED DESCRIPTION:
Primary treatment of clinical early-stage endometrial cancer consists of total hysterectomy, bilateral salpingo-oophorectomy, and lymph node assessment for staging. Sentinel lymph node (SLN) biopsy using indocyanine green (ICG) has been recommended in international guidelines as an alternative to systematic lymphadenectomy.

Conventional cervical ICG injection achieves bilateral SLN detection rates of approximately 73-75%. Re-injection may increase detection but prolongs the procedure. To optimize this approach, the investigators developed a modified technique in which ICG injection is continued until real-time lymphatic channels are visualized intraoperatively using the Firefly fluorescence mode of the robotic system.

The trial was designed as a prospective, randomized study comparing the conventional method with the modified technique in patients with clinical early-stage endometrial cancer undergoing robotic surgery. Participants were randomized in a 1:1 ratio to either the conventional cervical ICG injection group or the real-time lymphatic channel-guided ICG injection group. Randomization was performed using a computer-generated random sequence.

Initially, a sample size of 24 participants per group was planned, assuming bilateral detection rates of 75% (conventional) and 99% (modified). During the course of the study, the observed rates were 82.5% and 97.5%, respectively. A revised power analysis indicated the need for 40 participants per group, and the protocol was amended accordingly.

The study was completed with 40 participants in each group. The primary outcome was the rate of bilateral SLN detection. Secondary outcomes included operative parameters and perioperative complications.

ELIGIBILITY:
Inclusion Criteria: Patients with clinical stage 1-2 endometrial cancer ASA 1-3 patients. Ability to provide written informed consent

Exclusion Criteria: Patients with clinical stage 3-4 endometrial cancer Patients who are not suitable for robotic surgery due to their comorbidities (such as glaucoma, COPD, asthma) ASA 4-5 patients. Patients unable or unwilling to provide informed consent

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is limited to biologic females, as the study population is patients with endometrial cancer
Enrollment: 80 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Bilateral sentinel lymph node detection rate | Intraoperative (during surgery)
  Proportion of patients in whom sentinel lymph nodes are successfully identified bilaterally.

SECONDARY OUTCOMES:
Unilateral Sentinel Lymph Node Detection Rate | Intraoperative
  Proportion of patients in whom SLNs are detected unilaterally
Overall Sentinel Lymph Node Detection Rate (bilateral + unilateral) | Intraoperative
  Proportion of patients with any SLN detected
Operative Time | From skin incision to skin closure
  Total surgical duration measured in minutes
Time Required for Bilateral Sentinel Lymph Node Removal | Intraoperative (measured during surgery)
  The duration in minutes from the first cervical indocyanine green (ICG) injection to the successful removal of bilateral sentinel lymph nodes. This measure evaluates the efficiency of the mapping technique
Estimated Blood Loss | During surgery
  Amount of blood loss measured intraoperatively (mL)
Intraoperative and Postoperative Complications | Up to 30 days after surgery
  Any complications observed intraoperatively or within 30 days postoperatively

OTHER OUTCOMES:
Length of Hospital Stay | From immediately after surgery through hospital discharge (expected average of 2 days)
  Number of days from surgery to hospital discharge
Need for Blood Transfusion | Perioperative period
  Proportion of patients requiring intraoperative or postoperative blood product transfusion
Need for ICU Admission | From ICU admission through ICU discharge, an average of 1 day
  Proportion of patients requiring intensive care unit admission postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Gökhan Demirayak, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to patient privacy concerns and institutional regulations; however, de-identified aggregate data will be available upon reasonable request.

REFERENCES:
- [Result] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Result] 2- NCCN Clinical Practice Guidelines in Oncology. Uterine Neoplasms Version 4.2021 -September 3, 2021 https://www.nccn.org/professionals/physician_gls/pdf/uterine.pdf
- [Result] Yost KJ, Cheville AL, Al-Hilli MM, Mariani A, Barrette BA, McGree ME, Weaver AL, Dowdy SC. Lymphedema after surgery for endometrial cancer: prevalence, risk factors, and quality of life. Obstet Gynecol. 2014 Aug;124(2 Pt 1):307-315. doi: 10.1097/AOG.0000000000000372. PMID 25004343
- [Result] Maramai M, Achilarre MT, Aloisi A, Betella I, Bogliolo S, Garbi A, Maruccio M, Quatrale C, Aletti GD, Mariani A, Colombo N, Maggioni A, Multinu F, Zanagnolo V. Cervical re-injection of indocyanine green to improve sentinel lymph node detection in endometrial cancer. Gynecol Oncol. 2021 Jul;162(1):38-42. doi: 10.1016/j.ygyno.2021.04.026. Epub 2021 Apr 24. PMID 33906784